CLINICAL TRIAL: NCT06337357
Title: Evaluating Resistance Training for Sarcopenia in Older Patients With Type 2 Diabetes: Treatment Outcomes
Brief Title: Results of Progressive Resistance Training in Older Type 2 Diabetic Patients With Sarcopenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Geriatric Hospital (Other Government)
Responsible Party: Principal Investigator, Trinh Ngoc Anh, Endocrinologist, Principal Investigator and Sponsor, National Geriatric Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NatGerHos-Sarcopenia
Record Dates: First submitted 2024-03-13; First posted 2024-03-29 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia; Diabetes
Keywords: Sarcopenia; Diabetes; Resistance training
MeSH Terms: conditions — Sarcopenia; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group receives supervised resistance training instructions and baseline treatment for sarcopenia and diabetes:
  * Resistance training with elastic bands aims to increase muscle strength and muscle mass of the upper and lower limbs. Training duration 12 weeks, frequency 2 times/week, intensity gradually increases.
  * Baseline treatment for diabetes and sarcopenia: Recommendations according to American Diabetes Association guidelines which include instructions to follow the diet and exercises as recommended for older type 2 diabetic patients and baseline treatment for sarcopenia (education about sarcopenia and treatment measures such as diet and exercise) and provide basic information on resistance training.
  Interventions: Behavioral: Progressive Resistance Training
- Control group (No Intervention): The control group receives the baseline treatment for diabetes and sarcopenia:
  - Recommendations according to American Diabetes Association guidelines which include instructions to follow the diet and exercises as recommended for older type 2 diabetic patients and baseline treatment for sarcopenia (education about sarcopenia and treatment measures such as diet and exercise) and provide basic information on resistance training.

INTERVENTIONS:
Behavioral: Progressive Resistance Training — Progressive resistance training includes face-to-face education on resistance training:
  Resistance exercises with elastic bands include 9 exercises for 1 course. During the first 4 weeks, the patient exercises twice a week with a level of exertion according to Borg's category-ratio 10 (CR10) scale of 4-5 points. For the next 4 weeks, the patient exercises twice a week with Borg's CR10 exertion level of 6-7 points. In the last 4 weeks, the patient exercises twice a week with Borg's CR10 exertion level of 8-9 points.
  The three-month intervention involves twelve weekly calls, with a focus on building rapport (e.g. providing feedback on the baseline assessment); education reinforcement on resistance training; and skill-building (e.g. self-monitoring and resistance training diary). The emphasis is on helping participants to gain the knowledge and skills necessary to achieve targeted intensity. Every 4 weeks, all patients are re-visited by investigators in the hospital.
  Arms: Intervention group

SUMMARY:
A randomized controlled clinical trial that will test how progressive resistance training will impact outcomes of sarcopenia in older patients with type 2 diabetes who have been diagnosed as sarcopenia. The intervention will be 12 weeks in duration with approximately 24 sessions of resistance exercises. Outcome measures will be collected at baseline, 4, 8 weeks and 12 weeks.

DETAILED DESCRIPTION:
Sarcopenia, prevalent among geriatric populations, involves the progressive loss of muscle mass and decline in muscular function. This age-related condition is associated with higher susceptibility to falls, comorbidities, and mortality. Resistance training emerges as a non-pharmacological intervention proven to alleviate and potentially delay the progression of sarcopenia. However, there are still few studies investigating its effects on outcomes in older patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients diagnosed using American Diabetes Association 2022 criteria
* HbA1c ≥ 7.0 and ≤ 8.5%
* Sarcopenia diagnosed using criteria from the Asian Working Group for Sarcopenia 2019
* Age ≥ 60 and ≤ 80

Exclusion Criteria:

* Acute diabetic complications
* Patients are in the acute phase of musculoskeletal disorders: acute gout, progressing low-grade arthritis, acute joint pain due to joint degeneration, sciatic pain, and infectious arthritis.
* Patients suffer from conditions significantly affecting cognition and mobility: sequelae of stroke (with weakness, limb paralysis), muscular weakness, limb disabilities, severe heart failure, severe cognitive decline, and psychiatric disorders.
* Patients have been bedridden due to illness for more than 1 month within the past 3 months up to the recruitment time.
* Patients with cardiovascular diseases: chest pain, uncontrolled blood pressure ≥160/100 mmHg, untreated cardiac arrhythmia, a history of congestive heart failure, severe valvular heart disease, myocarditis or pericarditis, and hypertrophic cardiomyopathy.
* Renal failure with estimated glomerular function rate (Modification of Diet in Renal Disease equation) < 60 ml/min/m3 or serum creatinine ≥ 130 µmol/l
* On treatment with Sodium-glucose cotransporter 2 inhibitors (SGLT2i)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Physical performance 1 - Handgrip strength | Prior to the start of intervention, after 4 weeks, 8 weeks and 12 weeks (completion of the intervention)
  Handgrip strength is assessed using a hand dynamometer named Jamar Hydraulic Hand Dynamometer: the higher number the better outcome.
Physical performance 2 - Gait speed | Prior to the start of intervention, after 4 weeks, 8 weeks and 12 weeks (completion of the intervention)
  4-metre gait speed test (the shorter time the better outcome)
Physical performance 3 - Short Physical Performance Battery (SPPB) | Prior to the start of intervention, after 4 weeks, 8 weeks and 12 weeks (completion of the intervention)
  The Short Physical Performance Battery developed by the National Institute on Aging: scores ranging from 0 (worst) to 12 (best)
Muscle mass | Prior to the start of intervention, after 4 weeks, 8 weeks and 12 weeks (completion of the intervention)
  Upper and lower muscle mass are measured by Bioelectrical impedance analysis (BIA) method, using a machine model named InBody 770: the higher number the better outcome.

SECONDARY OUTCOMES:
Nutritional status | Prior to the start of intervention (Week 0), following the completion of the intervention (Week 12)
  Nutritional status is assessed using the Mini Nutritional Assessment Short-Form (MNA-SF): scores ranging from 0 (worst) to 14 (best)
Health-related Quality of Life | Prior to the start of intervention (Week 0), following the completion of the intervention (Week 12)
  Health-related Quality of Life is assessed using the health questionnaire 5-level 5 dimensions from EuroQol Group: index scores range from -0.59 to 1; 1 is the best possible health state.
Activities of Daily Living (ADLs) and Instrumental Activities of Daily Living (IADLs) | Prior to the start of intervention (Week 0), following the completion of the intervention (Week 12)
  Katz Index of Independence in Activities of Daily Living (scores range from 0-worst to 6-best) and Lawton Instrumental Activities of Daily Living Scale (scores range from 0-low function & dependent to 8-high function & independent for women, and 0-worst to 5-best for men)

CONTACTS AND LOCATIONS:
Overall Officials: Huyen TT Vu, PhD, Study Chair — National Geriatric Hospital
Locations (1):
- National Geriatric Hospital, Hanoi, Vietnam

REFERENCES:
- [Background] Mesinovic J, Zengin A, De Courten B, Ebeling PR, Scott D. Sarcopenia and type 2 diabetes mellitus: a bidirectional relationship. Diabetes Metab Syndr Obes. 2019 Jul 8;12:1057-1072. doi: 10.2147/DMSO.S186600. eCollection 2019. PMID 31372016
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Kerner W, Bruckel J; German Diabetes Association. Definition, classification and diagnosis of diabetes mellitus. Exp Clin Endocrinol Diabetes. 2014 Jul;122(7):384-6. doi: 10.1055/s-0034-1366278. Epub 2014 Jul 11. No abstract available. PMID 25014088
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Chen LK. The vicious cycle in the development of diabetes mellitus and sarcopenia in older persons. Arch Gerontol Geriatr. 2021 Jul-Aug;95:104437. doi: 10.1016/j.archger.2021.104437. Epub 2021 May 19. No abstract available. PMID 34029928
- [Background] Purnamasari D, Tetrasiwi EN, Kartiko GJ, Astrella C, Husam K, Laksmi PW. Sarcopenia and Chronic Complications of Type 2 Diabetes Mellitus. Rev Diabet Stud. 2022 Sep 28;18(3):157-165. doi: 10.1900/RDS.2022.18.157. PMID 36309772
- [Background] Chomentowski P, Coen PM, Radikova Z, Goodpaster BH, Toledo FG. Skeletal muscle mitochondria in insulin resistance: differences in intermyofibrillar versus subsarcolemmal subpopulations and relationship to metabolic flexibility. J Clin Endocrinol Metab. 2011 Feb;96(2):494-503. doi: 10.1210/jc.2010-0822. Epub 2010 Nov 24. PMID 21106709
- [Background] Russell ST, Rajani S, Dhadda RS, Tisdale MJ. Mechanism of induction of muscle protein loss by hyperglycaemia. Exp Cell Res. 2009 Jan 1;315(1):16-25. doi: 10.1016/j.yexcr.2008.10.002. Epub 2008 Oct 17. PMID 18973755
- [Background] Roubenoff R, Parise H, Payette HA, Abad LW, D'Agostino R, Jacques PF, Wilson PW, Dinarello CA, Harris TB. Cytokines, insulin-like growth factor 1, sarcopenia, and mortality in very old community-dwelling men and women: the Framingham Heart Study. Am J Med. 2003 Oct 15;115(6):429-35. doi: 10.1016/j.amjmed.2003.05.001. PMID 14563498
- [Background] Phillips T, Leeuwenburgh C. Muscle fiber specific apoptosis and TNF-alpha signaling in sarcopenia are attenuated by life-long calorie restriction. FASEB J. 2005 Apr;19(6):668-70. doi: 10.1096/fj.04-2870fje. Epub 2005 Jan 21. PMID 15665035
- [Background] Gobl C, Tura A. Focus on Nutritional Aspects of Sarcopenia in Diabetes: Current Evidence and Remarks for Future Research. Nutrients. 2022 Jan 13;14(2):312. doi: 10.3390/nu14020312. PMID 35057493
- [Background] Kumar P, Umakanth S, Girish N. A review of the components of exercise prescription for sarcopenic older adults. Eur Geriatr Med. 2022 Dec;13(6):1245-1280. doi: 10.1007/s41999-022-00693-7. Epub 2022 Sep 2. PMID 36050581
- [Background] Hurst C, Robinson SM, Witham MD, Dodds RM, Granic A, Buckland C, De Biase S, Finnegan S, Rochester L, Skelton DA, Sayer AA. Resistance exercise as a treatment for sarcopenia: prescription and delivery. Age Ageing. 2022 Feb 2;51(2):afac003. doi: 10.1093/ageing/afac003. PMID 35150587
- [Result] Ai Y, Xu R, Liu L. The prevalence and risk factors of sarcopenia in patients with type 2 diabetes mellitus: a systematic review and meta-analysis. Diabetol Metab Syndr. 2021 Sep 3;13(1):93. doi: 10.1186/s13098-021-00707-7. PMID 34479652
- [Result] Sanz-Canovas J, Lopez-Sampalo A, Cobos-Palacios L, Ricci M, Hernandez-Negrin H, Mancebo-Sevilla JJ, Alvarez-Recio E, Lopez-Carmona MD, Perez-Belmonte LM, Gomez-Huelgas R, Bernal-Lopez MR. Management of Type 2 Diabetes Mellitus in Elderly Patients with Frailty and/or Sarcopenia. Int J Environ Res Public Health. 2022 Jul 16;19(14):8677. doi: 10.3390/ijerph19148677. PMID 35886528
- [Result] Che S, Meng M, Jiang Y, Ye X, Xie C. Perceptions of exercise and exercise instruction in patients with type 2 diabetes mellitus and sarcopenia : a qualitative study. BMC Geriatr. 2022 Nov 22;22(1):892. doi: 10.1186/s12877-022-03519-0. PMID 36419014
- [Result] Studenski SA, Peters KW, Alley DE, Cawthon PM, McLean RR, Harris TB, Ferrucci L, Guralnik JM, Fragala MS, Kenny AM, Kiel DP, Kritchevsky SB, Shardell MD, Dam TT, Vassileva MT. The FNIH sarcopenia project: rationale, study description, conference recommendations, and final estimates. J Gerontol A Biol Sci Med Sci. 2014 May;69(5):547-58. doi: 10.1093/gerona/glu010. PMID 24737557
- [Result] Izzo A, Massimino E, Riccardi G, Della Pepa G. A Narrative Review on Sarcopenia in Type 2 Diabetes Mellitus: Prevalence and Associated Factors. Nutrients. 2021 Jan 9;13(1):183. doi: 10.3390/nu13010183. PMID 33435310
- [Result] Dai S, Shu D, Meng F, Chen Y, Wang J, Liu X, Xiao X, Guo W, Chen F. Higher Risk of Sarcopenia in Older Adults with Type 2 Diabetes: NHANES 1999-2018. Obes Facts. 2023;16(3):237-248. doi: 10.1159/000530241. Epub 2023 Apr 3. PMID 37011596
- [Result] Sugimoto K, Tabara Y, Ikegami H, Takata Y, Kamide K, Ikezoe T, Kiyoshige E, Makutani Y, Onuma H, Gondo Y, Ikebe K, Ichihashi N, Tsuboyama T, Matsuda F, Kohara K, Kabayama M, Fukuda M, Katsuya T, Osawa H, Hiromine Y, Rakugi H. Hyperglycemia in non-obese patients with type 2 diabetes is associated with low muscle mass: The Multicenter Study for Clarifying Evidence for Sarcopenia in Patients with Diabetes Mellitus. J Diabetes Investig. 2019 Nov;10(6):1471-1479. doi: 10.1111/jdi.13070. Epub 2019 Jun 1. PMID 31074209
- [Result] Chung SM, Moon JS, Chang MC. Prevalence of Sarcopenia and Its Association With Diabetes: A Meta-Analysis of Community-Dwelling Asian Population. Front Med (Lausanne). 2021 May 20;8:681232. doi: 10.3389/fmed.2021.681232. eCollection 2021. PMID 34095184
- [Result] Hong S, Chang Y, Jung HS, Yun KE, Shin H, Ryu S. Relative muscle mass and the risk of incident type 2 diabetes: A cohort study. PLoS One. 2017 Nov 30;12(11):e0188650. doi: 10.1371/journal.pone.0188650. eCollection 2017. PMID 29190709
- [Result] Wu H, Liu M, Chi VTQ, Wang J, Zhang Q, Liu L, Meng G, Yao Z, Bao X, Gu Y, Zhang S, Sun S, Zhou M, Jia Q, Song K, Huang J, Huo J, Zhang B, Ding G, Niu K. Handgrip strength is inversely associated with metabolic syndrome and its separate components in middle aged and older adults: a large-scale population-based study. Metabolism. 2019 Apr;93:61-67. doi: 10.1016/j.metabol.2019.01.011. Epub 2019 Jan 25. PMID 30690038
- [Result] Lee CG, Boyko EJ, Strotmeyer ES, Lewis CE, Cawthon PM, Hoffman AR, Everson-Rose SA, Barrett-Connor E, Orwoll ES; Osteoporotic Fractures in Men Study Research Group. Association between insulin resistance and lean mass loss and fat mass gain in older men without diabetes mellitus. J Am Geriatr Soc. 2011 Jul;59(7):1217-24. doi: 10.1111/j.1532-5415.2011.03472.x. Epub 2011 Jun 30. PMID 21718263
- [Result] Yang Q, Zhang Y, Zeng Q, Yang C, Shi J, Zhang C, Ni X, Du Z, Tang Z, Hu J, Li X, Cai J, Li Q, Cheng Q. Correlation Between Diabetic Peripheral Neuropathy and Sarcopenia in Patients with Type 2 Diabetes Mellitus and Diabetic Foot Disease: A Cross-Sectional Study. Diabetes Metab Syndr Obes. 2020 Feb 13;13:377-386. doi: 10.2147/DMSO.S237362. eCollection 2020. PMID 32104034
- [Result] Solerte SB, Gazzaruso C, Bonacasa R, Rondanelli M, Zamboni M, Basso C, Locatelli E, Schifino N, Giustina A, Fioravanti M. Nutritional supplements with oral amino acid mixtures increases whole-body lean mass and insulin sensitivity in elderly subjects with sarcopenia. Am J Cardiol. 2008 Jun 2;101(11A):69E-77E. doi: 10.1016/j.amjcard.2008.03.004. PMID 18514630
- [Result] Naseeb MA, Volpe SL. Protein and exercise in the prevention of sarcopenia and aging. Nutr Res. 2017 Apr;40:1-20. doi: 10.1016/j.nutres.2017.01.001. Epub 2017 Jan 16. PMID 28473056
- [Result] Martinez-Arnau FM, Fonfria-Vivas R, Cauli O. Beneficial Effects of Leucine Supplementation on Criteria for Sarcopenia: A Systematic Review. Nutrients. 2019 Oct 17;11(10):2504. doi: 10.3390/nu11102504. PMID 31627427
- [Result] Uchitomi R, Oyabu M, Kamei Y. Vitamin D and Sarcopenia: Potential of Vitamin D Supplementation in Sarcopenia Prevention and Treatment. Nutrients. 2020 Oct 19;12(10):3189. doi: 10.3390/nu12103189. PMID 33086536
- [Result] Beaudart C, Buckinx F, Rabenda V, Gillain S, Cavalier E, Slomian J, Petermans J, Reginster JY, Bruyere O. The effects of vitamin D on skeletal muscle strength, muscle mass, and muscle power: a systematic review and meta-analysis of randomized controlled trials. J Clin Endocrinol Metab. 2014 Nov;99(11):4336-45. doi: 10.1210/jc.2014-1742. Epub 2014 Jul 17. PMID 25033068
- [Result] Antoniak AE, Greig CA. The effect of combined resistance exercise training and vitamin D3 supplementation on musculoskeletal health and function in older adults: a systematic review and meta-analysis. BMJ Open. 2017 Jul 20;7(7):e014619. doi: 10.1136/bmjopen-2016-014619. PMID 28729308
- [Result] Gkekas NK, Anagnostis P, Paraschou V, Stamiris D, Dellis S, Kenanidis E, Potoupnis M, Tsiridis E, Goulis DG. The effect of vitamin D plus protein supplementation on sarcopenia: A systematic review and meta-analysis of randomized controlled trials. Maturitas. 2021 Mar;145:56-63. doi: 10.1016/j.maturitas.2021.01.002. Epub 2021 Jan 12. PMID 33541563
- [Result] Ganapathy A, Nieves JW. Nutrition and Sarcopenia-What Do We Know? Nutrients. 2020 Jun 11;12(6):1755. doi: 10.3390/nu12061755. PMID 32545408
- [Result] Krzyminska-Siemaszko R, Czepulis N, Lewandowicz M, Zasadzka E, Suwalska A, Witowski J, Wieczorowska-Tobis K. The Effect of a 12-Week Omega-3 Supplementation on Body Composition, Muscle Strength and Physical Performance in Elderly Individuals with Decreased Muscle Mass. Int J Environ Res Public Health. 2015 Aug 28;12(9):10558-74. doi: 10.3390/ijerph120910558. PMID 26343698
- [Result] Holten MK, Zacho M, Gaster M, Juel C, Wojtaszewski JF, Dela F. Strength training increases insulin-mediated glucose uptake, GLUT4 content, and insulin signaling in skeletal muscle in patients with type 2 diabetes. Diabetes. 2004 Feb;53(2):294-305. doi: 10.2337/diabetes.53.2.294. PMID 14747278
- [Result] Hovanec N, Sawant A, Overend TJ, Petrella RJ, Vandervoort AA. Resistance training and older adults with type 2 diabetes mellitus: strength of the evidence. J Aging Res. 2012;2012:284635. doi: 10.1155/2012/284635. Epub 2012 Sep 4. PMID 22988507
- [Result] Lee J, Kim D, Kim C. Resistance Training for Glycemic Control, Muscular Strength, and Lean Body Mass in Old Type 2 Diabetic Patients: A Meta-Analysis. Diabetes Ther. 2017 Jun;8(3):459-473. doi: 10.1007/s13300-017-0258-3. Epub 2017 Apr 5. PMID 28382531
- [Result] Zhang Y, Zou L, Chen ST, Bae JH, Kim DY, Liu X, Song W. Effects and Moderators of Exercise on Sarcopenic Components in Sarcopenic Elderly: A Systematic Review and Meta-Analysis. Front Med (Lausanne). 2021 May 19;8:649748. doi: 10.3389/fmed.2021.649748. eCollection 2021. PMID 34095166
- [Result] Yee XS, Ng YS, Allen JC, Latib A, Tay EL, Abu Bakar HM, Ho CYJ, Koh WCC, Kwek HHT, Tay L. Performance on sit-to-stand tests in relation to measures of functional fitness and sarcopenia diagnosis in community-dwelling older adults. Eur Rev Aging Phys Act. 2021 Jan 8;18(1):1. doi: 10.1186/s11556-020-00255-5. PMID 33419399
- [Result] Katula JA, Rejeski WJ, Marsh AP. Enhancing quality of life in older adults: a comparison of muscular strength and power training. Health Qual Life Outcomes. 2008 Jun 13;6:45. doi: 10.1186/1477-7525-6-45. PMID 18554394

DOCUMENTS (1):
  • Informed Consent Form (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT06337357/ICF_000.pdf